CLINICAL TRIAL: NCT01144130
Title: Postoperative Sleep Disturbances After Fast Track Hip and Knee Replacement
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lundbeck Center for Fast-Track Hip and Knee Replacement (Unknown)
Responsible Party: Lene Krenk, Doctor, Lundbeckcenter for fasttrack hip and knee replacement
Other Study IDs: H-2-2010-011
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2010-10

CONDITIONS: REM Sleep Measurement

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to quantify the degree of sleep disturbances after hip or knee replacement surgery.

Through polysomnographic monitoring the disturbances in sleep stages will be clarified.

ELIGIBILITY:
Inclusion Criteria:

* above 60
* ASA classification I-IV

Exclusion Criteria:

* general anaesthesia within 90 days
* daily use of sedatives
* alcohol abuse
* insufficient written and verbal Danish
* severe hearing loss and poor sight
* Parkinsons Disease or other functional neurological deficits
* Mini mental status < 24

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 60 years undergoing hip/knee replacement surgery in a fest track set-up.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Duration of REM sleep before and first postoperative night

CONTACTS AND LOCATIONS:
Overall Officials: Lene Krenk, Doctor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark